CLINICAL TRIAL: NCT01319149
Title: A Retrospective Study Of the Effects of Molecular Diagnostic Directed Wound Gels on Wound Care Outcomes
Brief Title: A Study of the Effects of Molecular Diagnostic Directed Wound Gels on Wound Care Outcomes
Status: Completed | Type: Observational
Sponsor: Southwest Regional Wound Care Center (Other)
Responsible Party: Principal Investigator, Randall Wolcott, Principal Investigator, Southwest Regional Wound Care Center
Other Study IDs: 56-RW-020
Record Dates: First submitted 2011-03-10; First posted 2011-03-21 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Wounds
Keywords: molecular methods
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: Patient records would be extracted from the electronic health record system of Southwest Regional Wound Care Center and placed in a separate bin.

SUMMARY:
A retrospective molecular diagnostic review on wound care outcomes. The time periods include March, April, May of 2010.The retrospective review would analyze the days of healing during the timeframe, upon the introduction of molecular diagnostic testing

DETAILED DESCRIPTION:
The null hypothesis would be that the introduction of molecular methods did not statistically affect patient outcomes. To study this hypothesis, our chief information technologist would query the database for any patients who are admitted during that time period. This period of time designated is March, April and May 2010.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been treated at SWRWCC during the months of March, April, or May 2010.

Exclusion Criteria:

* Patients who were not treated at SWRWCC during the time frame of March, April or May 2010.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with wounds who have been treated at Southwest Regional Wound Care Center.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The retrospective review would analyze the days of healing during the timeframe, upon the introduction of molecular diagnostic testing. | 1 yr
  To study this hypothesis, our chief information technologist would query the database for any patients who are admitted during that time period. This period of time designated is March, April and May 2010.

CONTACTS AND LOCATIONS:
Overall Officials: Randall D Wolcott, M.D., Principal Investigator — Southwest Regional Wound Care Center
Locations (1):
- Southwest Regional Wound Care Center, Lubbock, Texas, United States